CLINICAL TRIAL: NCT03642366
Title: Low-intensity Shockwaves Therapy Co-administered With Tadalafil 5mg for the Treatment of Severe, Vasculogenic Erectile Dysfunction:Validation of an Evidence Based Protocol in a Randomized, Sham-controlled Trial
Brief Title: Low-intensity Shockwaves Therapy + Tadalafil 5mg for the Treatment of Severe Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, Chairman, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10673/2018
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Erectile Dysfunction
Keywords: Low Intensity Shockwave Therapy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Arm 1 (Active Comparator)
  Interventions: Other: Dornier Aries2 LiST Device + 5mg Tadalafil (1)
- Active Arm 2 (Active Comparator)
  Interventions: Other: Dornier Aries2 LiST Device + 5mg Tadalafil (2)
- Sham Arm (Sham Comparator)
  Interventions: Other: Sham LiST Device + 5mg Tadalafil

INTERVENTIONS:
Other: Dornier Aries2 LiST Device + 5mg Tadalafil (1) — Patients will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), three times a week (total of 4 weeks) without treatment interval. Starting at first LiST session and finishing at the final week of LiST sessions, subjects will receive Tadalafil 5mg for 4 weeks daily. Total treatment period = 4 weeks.
  Arms: Active Arm 1
Other: Dornier Aries2 LiST Device + 5mg Tadalafil (2) — Patients will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), three times a week (total of 4 weeks) without treatment interval. Starting at first LiST session and finishing at the final week of LiST sessions, subjects will receive Tadalafil 5mg for 4 weeks daily. Total treatment period = 4 weeks.
  Arms: Active Arm 2
Other: Sham LiST Device + 5mg Tadalafil — Patients will receive sham shockwave treatment (12 sessions for all subjects, 5000 shockwaves at each session, at energy level 7)using a sham probe identical to active probes, three times a week (total of 4 weeks) without treatment interval. Starting at first LiST session and finishing at the final week of LiST sessions, subjects will receive Tadalafil 5mg for 4 weeks daily. Total treatment period = 4 weeks. The IIEF-ED domain will be evaluated at Visit 1 and, consequently, at baseline and all follow up visits together with the SEP diaries.
  Arms: Sham Arm

SUMMARY:
This is a randomized, double-blind, sham-controlled, 3 parallel arms, clinical trial. All patients will be PDE5I users or ex-users. After 1 month wash-out period, ED patients will be screened, in order to randomize 51 men with vasculogenic ED. Patients will be randomized in 3 groups (17 subjects in each group) to receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), three times a week (total of 4 weeks) without treatment interval. One group will be sham-control at energy level 7 whereas 2 groups will receive active treatment.Three identical standard probes (probes A, B, C) will be used for the study, 2 of them active and one sham. Starting at first LiST session and finishing at the final week of LiST sessions, subjects will receive Tadalafil 5mg for 4 weeks daily. Total treatment period = 4 weeks. The IIEF-ED domain will be evaluated at Visit 1 and, consequently, at baseline and all follow up visits together with the SEP diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 40-70 years.
3. Sexually active in a stable, heterosexual relationship of more than three months duration.
4. Presence of Erectile Dysfunction for at least 6 months.
5. At screening, diagnosed as Vasculogenic erectile dysfunction based on sexual history.
6. Partial response to highest dose of PDE5i
7. Agree to suspend all other ED therapies, except the assigned study treatments, for the duration of the study.
8. Agree to attempt sexual intercourse and document the outcome using the Sexual Encounter Profile (SEP) at least 4 times for the last 4 weeks prior to Visit 2/Randomization, 1 month Follow Up, 3 month Follow Up and 4 month Follow Up without being under the influence of alcohol or recreational drugs. Agree to document the outcome using the Sexual Encounter Profile (SEP) diary.
9. IIEF-ED score 1-10 at Visit 2 (after PDE5i washout)
10. At Visit 2 (after PDE5i washout), SEP Q2, "Were you able to insert your penis into your partner's vagina?" answered "YES" 0 - 50% of the time.
11. At Visit 2, SEP Q3, "Did your erection last long enough for you to have successful intercourse?" answered "YES" 0 - 25% of the time.

Exclusion Criteria:

1. Previous major pelvic surgery or pelvic trauma that could impact erectile function, such as radical prostatectomy, radical cystectomy, rectal surgery. Patients with previous TURP surgery without sequelae of iatrogenic ED may be included.
2. Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, grafting.
3. Previous history of priapism or penile fracture
4. Previous radiation therapy to pelvis.
5. Abnormal serum testosterone level defined as a value lower than 300 ng/dL (indicative of untreated hypogonadism), or greater than 1197 ng/dL.
6. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
7. ED due primarily to psychogenic factors.
8. Peyronie's Disease or penile curvature that negatively influences sexual activity.
9. Patients with cardiac or non-cardiac electrical devices implanted.
10. Open wound or any anatomical or neurological abnormalities in the treatment area.
11. Uncontrolled diabetes mellitus with glucose >200 mg/dL (once or more times/week during the last month prior to recruitment, or during screening blood test).
12. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson 's disease.
13. Refusal to suspend ED therapy for duration of study. Subjects who are using Tadalafil as a treatment for BPH (Benign Prostatic Hyperplasia) will also be excluded.
14. Men deemed not healthy enough to participate in sexual activity.
15. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
16. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
17. Known allergy to ultrasound gel. 18,. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using SSRI or psychotropic medications e.g., Citalopram (Celexa), Escitalopram (Lexapro, Cipralex), Paroxetine (Paxil, Seroxat), Fluoxetine (Prozac), Fluvoxamine (Luvox, Faverin),Sertraline (Zoloft, Lustral), Clonazepam (Klonopin), Alprazolam (Xanax), Aripiprazole (Ambilify), Clozapine (Clozaril), Risperidone (Risperdal), Quetiapine (Seroquel), Olanzapine (Zyprexa) are also excluded.

19. Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.

20. History of adverse events in response to tadalafil, which would prevent patient compliance to the study protocol.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The difference between the groups in the change of the Erectile Function (EF) domain score of the International Index of Erectile (IIEF) | baseline and 12 week follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)

SECONDARY OUTCOMES:
The difference between the groups in the change of the Erectile Function (EF) domain score of the International Index of Erectile (IIEF) | baseline and 4 week follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
The difference between the groups in the change of the Erectile Function (EF) domain score of the International Index of Erectile (IIEF) | baseline and 16 week follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 4-week follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 12-week follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 16-week follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Number of patients with treatment related adverse events | 20 weeks
  Potential treatment related adverse events after the first LI-ESWT session and during the 16-weeks follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases, Thessaloniki, Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece